CLINICAL TRIAL: NCT06260475
Title: IUA Committee Research Project on the Management of TASC C and D Aortoiliac Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Clinical Centre of Serbia (Other); University of Padova (Other); University of Bari (Other); University of Trieste (Other); University of Nis (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro (Other); Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, Clinical Professor, Universidade do Porto
Other Study IDs: IUA - 246-18
Record Dates: First submitted 2023-12-10; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Aortoiliac Atherosclerosis; Aortoiliac Occlusive Disease; Aortoiliac Atherosclerosis With Gangrene; Aortoiliac Atherosclerosis Without Gangrene; Aortoiliac Obstruction; Peripheral Arterial Disease; Peripheral Vascular Diseases
Keywords: peripheral artery disease;; aortobifemoral bypass;; aortoiliac stenting;; preoperative care;
MeSH Terms: conditions — Leriche Syndrome; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with symptomatic peripheral artery disease and aortoiliac obstrutive disease: Chronic limb-threatening ischemia or claudicants due to extensive Aortoiliac Occlusive Disease (AIOD), particularly in Trans-Atlantic Inter-Society Consensus II (TASC-II) type C and D lesions
  Interventions: Procedure: Aortobifemoral bypass; Procedure: aortoiliac stenting

INTERVENTIONS:
Procedure: Aortobifemoral bypass — Open surgery with aortic and iliac reconstruction
  Other Names: aortobiliac bypass
Procedure: aortoiliac stenting — Endovascular reconstruction of aortic and iliac arterial obstruction:
  Balloon angioplasty may be performed initially to dilate the narrowed segment of the iliac artery.
  Subsequently, a stent delivery system is advanced over the wire and positioned across the lesion.
  The stent is deployed under fluoroscopic guidance to expand and scaffold the diseased artery, restoring blood flow.
  Vascular - iliac dedicated Stent - any brand
  Other Names: Percutaneous transluminal aortoiliac stenting; Endovascular treatment of aortoiliac occlusive disease

SUMMARY:
This study aims to evaluate the clinical, imaging results of endovascular revascularization of the aorto-iliac sector in comparison with aortobifemoral bypass and the hybrid approach, in patients with atherosclerotic disease of the iliac sector classified as type C and D by the TransAtlantic Inter-Society Consensus (TASC II

DETAILED DESCRIPTION:
Open surgery repair with Aortobifemoral Bypass (ABF) remains the gold standard revascularization technique in patients with lifestyle-limiting intermittent claudication (IC) and chronic limb-threatening ischemia due to extensive Aortoiliac Occlusive Disease (AIOD), particularly in Trans-Atlantic Inter-Society Consensus II (TASC-II) type D lesions

The ABF procedure has proven safe, effective, and durable, particularly considering its high long-term patency rates (85%-90% at five years and 75%-80% at ten years) despite its significant peri-operative associated morbidity (1). On the other hand, endovascular treatment (EVT) offers an attractive alternative with durable results (four- or 5-year primary and secondary patency rates ranged from 60% to 86% and 80% to 98%, respectively), especially in less extensive AIOD, while also providing less perioperative morbidity, making it generally preferable for patients with more severe comorbid conditions.

Thus, surgical approaches to extensive AIOD have changed considerably over the last years, primarily due to increased EVT, particularly with the uncovered aortoiliac stenting (AIS). While TASC II provides an anatomical framework to compare therapeutic techniques, the advancement of endovascular techniques has led to many trials suggesting that endovascular management of TASC II C and D lesions is a potential alternative treatment to open strategies. It is attractive for patients with high surgical risk, given the substantially less perioperative morbidity and mortality compared to ABF

This study aims to evaluate the clinical, imaging results of endovascular revascularization of the aorto-iliac sector in comparison with aortobifemoral bypass and the hybrid approach, in patients with atherosclerotic disease of the iliac sector classified as type C and D by the TransAtlantic Inter-Society Consensus (TASC II).

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial/atherosclerotic disease of the aorto-iliac sector undergoing direct, hybrid or endovascular surgical correction with TransAtlantic Inter-Society Consensus (TASC II) type D classification(12).

  * Age >18 years old

Exclusion Criteria:

* Synchronous aortoiliac aneurysmatic/ectasic disease (aorta AP diameter >25 mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revascularization of the aorto-iliac sector for peripheral arterial disease at any of the center in study starting in January 2016 until December 2023.A consecutive sample will be prepared, containing all patients at the recruiting centers, fulfilling the following criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Amputation | through study completion, an average of 3 years
  Amputation above the ankle
Cardiovascular Death | through study completion, an average of 3 years
  Death from cardiovascular disease
acute myorcardial infartion | through study completion, an average of 3 years
  According to the 4th definition of Myocardial infarction

SECONDARY OUTCOMES:
Major Adverse Limb Events | through study completion, an average of 3 years
  Amputation above the ankle, arterial thrombosis of the limb, binary restenosis
Major adverse cardiovascular events | through study completion, an average of 3 years
  acute myocardial infarction; acute heart faillure, cardiovascular death, coronary reintervention
Death | through study completion, an average of 3 years
  Diagnosed by a physician

OTHER OUTCOMES:
Intensive care unit instay | until 30 days
  Intensive care unit instay - days)
acute kidney injury (AKI) | until 30 days
  AKI according to Riffle criteria

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Centro Hospitalar Universitário de São João, EPE, Porto
  - Faculdade de Medicina da Universidade do Porto, Porto

IPD SHARING:
Plan to Share IPD: No
The anonymity and confidentiality of participants will be safeguarded. The patient will be entered without any reference to their name. The participant number will correspond to the clinical information in a separate database, which will only be used for the proposed objective after supervision by the PI and Supervisor. For analysis purposes, the participant number will be deleted.
  All information entered in the database will be constant in the clinical process.
  The results may be published in a scientific journal and/or congress. Rules of Ethical Conduct and Good Practices will be observed to ensure compliance with the precepts of the Declaration of Helsinki, the Convention on Human Rights and Biomedicine, the guidelines of the Council for International Organizations of Medical Sciences and the Guide to Good Clinical Practices.

REFERENCES:
- [Background] Jongkind V, Akkersdijk GJ, Yeung KK, Wisselink W. A systematic review of endovascular treatment of extensive aortoiliac occlusive disease. J Vasc Surg. 2010 Nov;52(5):1376-83. doi: 10.1016/j.jvs.2010.04.080. PMID 20598474
- [Background] Groot Jebbink E, Holewijn S, Slump CH, Lardenoije JW, Reijnen MMPJ. Systematic Review of Results of Kissing Stents in the Treatment of Aortoiliac Occlusive Disease. Ann Vasc Surg. 2017 Jul;42:328-336. doi: 10.1016/j.avsg.2017.01.009. Epub 2017 Apr 6. PMID 28390920